CLINICAL TRIAL: NCT04415216
Title: Long-term Outcomes Following Drug Eluting Balloon Versus Thin Struts Drug Eluting Stents for Treating In-stent Restenosis: Propensity Score-matched Analysis(DEB-Dragon Registry).
Brief Title: DEB vs Thin-DES in DES-ISR: Long Term Outcomes (DEB Dragon Registry)
Acronym: DEB-DRAGON
Status: Completed | Type: Observational
Sponsor: Medical University of Silesia (Other)
Collaborators: Wojciech Wojakowski (Unknown)
Responsible Party: Principal Investigator, Wojciech Wańha, MD, PhD, Medical University of Silesia
Other Study IDs: 02
Record Dates: First submitted 2020-05-31; First posted 2020-06-04 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: In Stent Restenosis
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ISR PCI with thin-DES
  Interventions: Device: percutaneous coronary intervention
- ISR PCI with DEB
  Interventions: Device: percutaneous coronary intervention

INTERVENTIONS:
Device: percutaneous coronary intervention — Percutaneous coronary intervention with drug eluting balloon (DEB) vs. thin struts drug eluting stents (thin-DES) for treating in-stent restenosis (ISR)

SUMMARY:
Data regarding the usefulness of percutaneous coronary intervention (PCI) with drug eluting balloon (DEB) vs. thin struts drug eluting stents (thin-DES) for treating in-stent restenosis (ISR) in every day clinical practice is scarce. We aimed to evaluate comparing the efficacy and safety profile of DEB and thin-DES in DES-ISR.

ELIGIBILITY:
Inclusion Criteria:

• All consecutive patients with DES-ISR who were treated with either paclitaxel-DEB or thin-DES.

Exclusion Criteria:

* PCI with DES struts thickness >100μm
* PCI with DEB and thin-DES in the same procedure
* PCI of other vascular territories during the same procedure
* PCI in saphenous vain graft or internal mammary artery

Age Groups: Child, Adult, Older Adult
Study Population: Patients with DES-ISR who were treated with either paclitaxel-DEB or thin-DES
Sampling Method: Probability Sample
Enrollment: 1369 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
TLR | 3 years
  target lesion revascularisation

SECONDARY OUTCOMES:
DOCE | 3 years
  composite of cardiac death, TLR, and target vessel MI
TVR | 3 years
  target vessel revascularization
TV-MI | 3 years
  target vessel myocardial infarction
cardiac death | 3 years
myocardial infarction | 3 years

CONTACTS AND LOCATIONS:
Locations (9):
- Poland (9):
  - Department of Invasive Cardiology, Medical University of Bialystok, Bialystok
  - Cardiovascular Institute, Nicolaus Copernicus University, Bydgoszcz, Poland, Bydgoszcz
  - First Department of Cardiology, Medical University of Gdansk, Gdansk, Poland, Gdansk
  - Department of Cardiology and Structural Heart Diseases, Medical University of Silesia, Katowice, Poland, Katowice
  - Second Department of Cardiology, Jagiellonian University Medical College, Krakow, Poland, Krakow
  - Department of Interventional Cardiology and Angiology, National Institute of Cardiology, Warsaw, Poland, Warsaw
  - Department of Invasive Cardiology, Centre of Postgraduate Medical Education, Central Clinical Hospital of the Ministry of Interior and Administration, Warsaw
  - Centre for Heart Disease, University Hospital Wroclaw Department of Heart Disease, Wroclaw Medical University, Wroclaw
  - Third Department of Cardiology, Medical University of Katowice, Zabrze

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] De Filippo O, Wanha W, Sanavia T, Januszek R, Giacobbe F, Campo G, Pinxterhuis TH, Capodanno D, Tomasiewicz B, Iannaccone M, Leone A, Wolny R, Bruno F, Patti G, Musumeci G, Liccardo G, Verardi R, Roubin SR, Tarantini G, Kuzma L, Perl L, Gagnor A, Reczuch K, Conrotto F, Tuttolomondo D, Ploumen EH, Niezgoda P, Caglioni S, Omede P, Greco A, Kubica J, Gil RJ, Piccolo R, Kornowski R, Bil J, Morena A, Zocca P, Pennone M, Gasior M, Jaguszewski M, von Birgelen C, Fariselli P, De Ferrari GM, Wojakowski W, D'Ascenzo F. Treatment of in-stent restenosis with ultrathin-strut versus thin-strut drug-eluting stents or drug-eluting balloons: a multicentre registry. EuroIntervention. 2024 Nov 4;20(21):e1340-e1354. doi: 10.4244/EIJ-D-24-00491. PMID 39492702
- [Derived] Wanha W, Bil J, Januszek R, Gilis-Malinowska N, Figatowski T, Milewski M, Pawlik A, Staszczak B, Wybraniec M, Tomasiewicz B, Kubler P, Kuliczkowski W, Walczak T, Hrymniak B, Desperak P, Mielczarek M, Ciecwierz D, Niezgoda P, Wolny R, Chudzik M, Kuzma L, Kralisz P, Kedhi E, D'Ascenzo F, Hudziak D, Kowalowka A, Smolka G, Reczuch K, Gruchala M, Kubica J, Gil RJ, Dobrzycki S, Dudek D, Bartus S, Gasior M, Ochala A, Witkowski A, Jaguszewski M, Wojakowski W. Long-Term Outcomes Following Drug-Eluting Balloons Versus Thin-Strut Drug-Eluting Stents for Treatment of In-Stent Restenosis (DEB-Dragon-Registry). Circ Cardiovasc Interv. 2021 Sep;14(9):e010868. doi: 10.1161/CIRCINTERVENTIONS.121.010868. Epub 2021 Sep 3. PMID 34474584